CLINICAL TRIAL: NCT02843360
Title: National Health Interview Survey in Taiwan
Acronym: NHIS
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: NHISTaiwan
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Public Health
Keywords: public health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The major elements of the survey were sampling, questionnaire design, field survey and database construction. This survey incorporated the multistage stratified sampling scheme. Questionnaires include health status, utilization of health care, health behaviors, quality of life, and social economic status.

DETAILED DESCRIPTION:
This survey took a representative sample from each county and municipality in Taiwan using a stratified multi-stage systematic sampling procedure. Within each county/municipality (stratum), samples were selected with probability proportional to population size. Questionnaire design was based on the needs of the Department of Health and Welfare and the public health professionals. Due to different age has different health problems, the questionnaires were divided into 3 parts: under 12, 23-64, and 65+ years. The response rate was 75% in 2013.

ELIGIBILITY:
Inclusion Criteria:

* All the selected samples were to be interviewed.

Exclusion Criteria:

* severely ill or too frail to answer;
* having cognitive problems;
* having hearing or speaking problems; or
* dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the community dwelling people were eligible for the survey.
Sampling Method: Probability Sample
Enrollment: 23296 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Health Status of the General Population | 1 year
  Survey on the general health of the nation in a specific time

IPD SHARING:
Plan to Share IPD: No